CLINICAL TRIAL: NCT01275430
Title: A Study to Assess the Precision of the Sherlock 3CG Tip Positioning System as a Tool to Guide Peripherally Inserted Central Catheter Placement
Brief Title: Assessment of the Precision of the Sherlock 3CG Tip Positioning System
Acronym: STAT-PICC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Phase I completed. Phase II is cancelled.
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BAS-3004
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Results first posted 2016-07-04 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: No Specific Conditions Under Study. Primary Focus: Adult Subjects Who Require PICC Placement
Keywords: central venous catheters; peripherally inserted central catheters (PICC_; Electrocardiography (ECG); intravascular ECG; Tip Positioning System

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sherlock 3CG (Experimental): Sherlock 3CG is indicated for central venous catheter guidance and positioning during catheter placement. The Sherlock 3CG provides real time catheter tip location information through the use of passive magnet and cardiac electrical signal detection.
  Interventions: Device: Sherlock 3CG
- "Blind" Placement (Active Comparator): PICCs will be placed "blindly", without the use of any tip location/positioning device.
  Interventions: Other: Blind Placement

INTERVENTIONS:
Device: Sherlock 3CG — Sherlock 3CG is indicated for central venous catheter guidance and positioning during catheter placement. The Sherlock 3CG provides real time catheter tip location information through the use of passive magnet and cardiac electrical signal detection.
  Arms: Sherlock 3CG
Other: Blind Placement — PICCs will be placed "blindly", without the use of any tip location/positioning device.
  Arms: "Blind" Placement

SUMMARY:
Phase I

* determine the location of the peripherally inserted central catheter (PICC) tip upon observation of maximum p-wave amplitude

Phase II

* determine the precision of PICC placement in the Sherlock 3CG group versus the standard PICC placement

DETAILED DESCRIPTION:
The feasibility phase of this study (Phase I) is a prospective, single arm, single-center feasibility study to determine the distance of the PICC tip to the upper Caval Atrial junction upon observation of maximum p-wave after PICC tip placement using the Sherlock 3CG system. Subjects judged by site personnel to require PICC placement will be screened against the study inclusion/exclusion criteria. Those subjects meeting the study criteria will be offered enrollment into the study. Informed consent will be obtained prior to subject enrollment.

PICC nurses who have been fully trained in the correct use of the Sherlock 3CG Tip Positioning System will perform the PICC placement procedures in the fluoroscopy suite. Serious adverse events (SAEs) will be collected, but collection of non-serious AEs will be limited to those adverse events (AEs) considered to be study procedure and/or device-related.

Subject follow up will be complete 30 days following the date of the study PICC procedure.

The results of the feasibility phase will be used to determine:

1. the distance, if any, that is required to move the PICC tip upon observation of the maximum p-wave amplitude in the pivotal phase of the study (See Section 3.5.3), in order to have the PICC tip at the upper cavoatrial junction.
2. the movement of the cardiovascular anatomy, if any, when the arm is adducted from above the head to the side of the subject.
3. the movement of the PICC tip when the arm is moved from the 90° angle to the side.

Phase II (Pivotal) will not begin until the Phase I (feasibility) is complete. The Phase II study is a prospective, single-center, controlled, blinded, randomized study to compare the Sherlock 3CG as a tool in guiding PICC placement to the standard "blind" technique (control). Subjects judged by site personnel to require PICC placement will be screened against the study inclusion/exclusion criteria. Those subjects meeting the study criteria will be offered participation into the study. Informed consent will be obtained prior to subject enrollment. Subjects will be randomly assigned to either the Sherlock 3CG group or the control group in a 1:1 fashion. Due to the different placement techniques being utilized, the PICC nurses and study coordinator will not be blinded to the study device. PICC nurses who have been fully trained in the correct use of the Sherlock 3CG will perform the PICC placement procedures in the fluoroscopy suite. Serious adverse events (SAEs) will be collected, but collection of non-serious AEs will be limited to those AEs considered to be study procedure and/or device-related. Subject follow up will be complete 30 days following the date of the study PICC procedure.

Randomization did not occur due to early termination. All participants were assigned to Sherlock 3CG in phase I. Randomization would have occurred at the start of Phase II, but Phase II was not initiated due to early termination. Phase II was cancelled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 21years
2. Require 5 F dual lumen or 4 F single lumen PowerPICC or PowerPICC SOLO placement as part of standard care
3. Be able to undergo study procedures
4. Subject is able to comply with all study requirements and be available for 30 day follow-up visit.
5. Subject has signed an Informed Consent Form (ICF) or has had an ICF signed by the subject's legally authorized representative

Exclusion Criteria:

1. Subject has a contraindication to PICC placement as listed in the Instructions for Use (IFU) (See Section 18.2)
2. Subject has been previously randomized for this study.
3. Subject is unable to lie in the supine position on the fluoroscopy table
4. Subject had radiation therapy within the last three years
5. Subject has an existing pregnancy
6. Subject has known glomerular filtration rate (GFR) <45 ml/min/1.73m2
7. Subject has a functioning pacemaker or defibrillator
8. Subject has an artificial heart or heart transplant
9. Subject has anatomical abnormalities of the central venous system
10. Subject has atrial fibrillation or other atrial arrhythmias in which a p-wave was not consistently present on ECG
11. Subject has internal wires that may interfere with imaging
12. Subject has an existing central venous catheter
13. Subject is unable to raise arms above the head while lying down.
14. Subject has a BMI ≥45
15. The clinician is unable to obtain accurate external measurement due to anatomical abnormalities or personal/medical equipment.
16. Subject has a known allergy or hypersensitivity to contrast media.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon McLennan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Phase I was feasibility and wasn't powered. Phase II was powered, but cancelled due to slow enrollment during Phase I.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sherlock 3CG: Subjects undergoing PICC placement had their PICCs placed in conjunction with the Sherlock 3CG Tip Confirmation System.
  All participants were assigned to Sherlock 3CG in Phase I. Zero subjects started Phase II because of early termination of the study, so zero subjects were randomized. All adverse event reporting is also for Phase I (3CG) participants.
Period: Overall Study
Arm/Group | Sherlock 3CG
Started | 27
Completed | 18
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — No Contrast Injection | 6
Not completed — Device Malfunction | 1
Not completed — Inability to achieve maximum p-wave | 1

BASELINE CHARACTERISTICS:
Population: Subjects undergoing PICC placement for long term IV therapy
Groups:
- Sherlock 3CG: Sherlock 3CG is indicated for central venous catheter guidance and positioning during catheter placement. The Sherlock 3CG provides real time catheter tip location information through the use of passive magnet and cardiac electrical signal detection.
  Randomization did not occur due to early termination. All participants were assigned to Sherlock 3CG in phase I. Randomization would have occurred at the start of Phase II, but Phase II was not initiated due to early termination.
Arm/Group | Sherlock 3CG
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13.2)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
Region of Enrollment [Number; unit: participants]
  United States | 18
Reason For PICC Placement [Number; unit: participants]
  Antibiotics | 17
  Total Parenteral Nutrition (TPN) | 1
Access Vein [Number; unit: participants]
  Brachial | 9
  Basilic | 9
Access Side [Number; unit: participants]
  Left | 6
  Right | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Location of the PICC Tip Upon Observation of Maximum P-wave Amplitude Using Sherlock 3CG.
Description: Mean distance (mm) from the PICC tip to the upper cavoatrial junction (CAJ) upon observation of maximum p-wave amplitude when using Sherlock 3CG.
  All subjects were assigned to Sherlock 3CG in Phase I. Randomization was to have occurred in Phase II, but Phase II was not initiated due to termination of the study.
Time Frame: Time of PICC placement (Day 0)
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Sherlock 3CG: Mean distance (mm) from the PICC tip to the upper Caval Atrial junction upon observation of maximum p-wave amplitude when using Sherlock 3CG.
Arm/Group | Sherlock 3CG
Number analyzed (Participants) | 18
mm
  PICC tip above upper CAJ | 18.8 (18.1)
  PICC tip below upper CAJ | 14.3 (10.0)

2. Secondary Outcome: Phase I: Distance Necessary for Repositioning of the PICC Tip Upon Observation of the Maximum P-wave Amplitude, if Necessary.
Description: Distance (mm), if any, that is required to move the PICC tip upon observation of the maximum p-wave amplitude in order to have the PICC tip at the upper cavoatrial junction. Direct measurement of distance from the catheter tips to the parts of the CAJ
  All subjects were assigned to Sherlock 3CG in Phase I. Randomization was to have occurred in Phase II, but Phase II was not initiated due to termination of the study.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Sherlock 3CG: Subjects undergoing PICC placement had their PICCs placed in conjunction with the Sherlock 3CG Tip Confirmation System
Arm/Group | Sherlock 3CG
Number analyzed (Participants) | 18
mm | 13.8 (2.0)

3. Secondary Outcome: Number of Participants With Acceptable Angiographic CT Visualization of the PICC Tip When Using Sherlock 3CG for PICC Placement
Description: Proportion of acceptable visualization of the PICC tip location when maximum p-wave amplitude is observed.
  Note - this endpoint is to assess the diagnostic capability of Angiographic Computed Tomography (ACT). It is not designed to reflect on PICC tip location.
  All subjects were assigned to Sherlock 3CG in Phase I. Randomization was to have occurred in Phase II, but Phase II was not initiated due to termination of the study.
Time Frame: Day 0
Measure: Number; unit: participants
Arm/Group | Sherlock 3CG
Number analyzed (Participants) | 18
participants | 18

4. Secondary Outcome: Phase I: Change in Distance (mm) Between the Location of the Cavoatrial Junction When Angiographic CT is Performed With the Arms Above the Head vs at the Subject's Side.
Description: Measurements (mm) of the location of the cavoatrial junction on Angiographic CT to evaluate shift greater than 5mm in mediastinal structures between ACT acquisitions obtained with the arms above the head vs arms at side of body (90°).
  All subjects were assigned to Sherlock 3CG in Phase I. Randomization was to have occurred in Phase II, but Phase II was not initiated due to termination of the study.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sherlock 3CG
Number analyzed (Participants) | 18
mm | 0 (0)

5. Secondary Outcome: Phase I: Amount of PICC Tip Movement When the Subject's Arm is Adducted From a 90° Position to the Subject's Side.
Description: Mean distance (mm) of PICC tip movement when the subject's arm is adducted from a 90° position to the subject's side, by directly measuring the distance from the catheter tips to the parts of the CAJ (upper, middle, and lower) with the subject's arm at 90°and compared to the PICC tip with the subject's arm at the side .
  All subjects were assigned to Sherlock 3CG in Phase I. Randomization was to have occurred in Phase II, but Phase II was not initiated due to termination of the study.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sherlock 3CG
Number analyzed (Participants) | 18
mm
  PICC tip moved caudally | 22.3 (12.0)
  PICC tip moved cephalad | 8.7 (7.0)

ADVERSE EVENTS:
Time Frame: 30 days following PICC placement procedure
Groups:
- Sherlock 3CG: Subjects undergoing PICC placement had their PICCs placed in conjunction with the Sherlock 3CG Tip Confirmation System
  All subjects were assigned to Sherlock 3CG in Phase I. Randomization was to have occurred in Phase II, but Phase II was not initiated due to termination of the study.
Arm/Group | Sherlock 3CG
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sherlock 3CG (N=27)
Extravasation (Surgical and medical procedures) | 1 — Subject had injection site extravasation. Subject recovered without sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No